CLINICAL TRIAL: NCT04187508
Title: A Phase IIa, Double-Blind, Randomized, Parallel Group, Placebo-Controlled Multi-Centre Study to Evaluate the Effect of AZD8154 Administered Via Nebulizer Once Daily on Allergen-Induced Inflammation in Subjects With Mild Allergic Asthma Challenged With an Inhaled Allergen
Brief Title: A Study to Evaluate the Effect of AZD8154 Administered Via Nebulizer Once Daily in Subjects With Mild Allergic Asthma Challenged With an Inhaled Allergen
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The reason is: emerging pre-clinical toxicology findings.
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D8900C00004
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Asthma
Keywords: Allergen-induced inflammation
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The study will be randomized and double blinded, ie, subjects, Investigators, and other study site personnel must be kept blinded to avoid bias, although due to the differences between the AZD8154 and placebo treatments unblinded pharmacy/site staff will be required for dose preparation and administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AZD8154 (Experimental): Subjects will receive AZD8154 QD dosing for 10 days
  Interventions: Drug: AZD8154 nebulizer suspension, 20 mg/mL
- Placebo (Placebo Comparator): Subjects will receive AZD8154 matching placebo QD dosing for 10 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD8154 nebulizer suspension, 20 mg/mL — Subjects will receive AZD8154 from Day 1 to Day 10 (10 consecutive days) by using nebulizer and dosimeter system as inhaled dosing and delivered dose will be 3mg.
  Arms: AZD8154
Drug: Placebo — Subjects will receive AZD8154 matching placebo (placebo nebulizer suspension, glucose solution for infusion 50 mg/mL) QD from Day 1 to Day 10 (10 consecutive days) by using nebulizer and dosimeter system as inhaled dosing.
  Arms: Placebo

SUMMARY:
This is a Phase IIa, double blind, randomized, parallel group, placebo controlled multi centre study to evaluate the effect of AZD8154 (administered via nebulizer daily [QD]) on allergen-induced inflammation in subjects with mild allergic asthma challenged with an inhaled allergen. Approximately 36 subjects who meet all eligibility criteria will be randomized (1:1) to receive either AZD8154 or placebo.

DETAILED DESCRIPTION:
This is a Phase IIa, double blind, randomized, parallel group, placebo controlled multi centre study which will include 36 subjects in total and 18 subjects in each treatment group are needed for this study.

AZD8154 or placebo is administered via nebulizer QD for 10 consecutive days. This study will include 5 sites in the AllerGen Clinical Investigator Collaborative (CIC) group in Canada.

ELIGIBILITY:
Inclusion Criteria:

Informed consent

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this Clinical Study Protocol (CSP).
* Provision of signed and dated, written ICF prior to any mandatory study specific procedures, sampling, and analyses.
* Provision of signed and dated written Genetic ICF prior to collection of samples for genetic analysis (if subject agrees to take part in this optional assessment).

Age • Subject must be 18 to 65 years of age (inclusive) at the time of signing the ICF.

Type of subject and disease characteristics

* Individuals who are determined as healthy by the Investigator, based on medical evaluations including, but not limited to, medical history, physical examination, laboratory tests, vital signs, and electrocardiogram (ECG).
* Subjects have mild, stable, allergic asthma with episodic wheeze and shortness of breath. Asthma therapy is limited to inhaled, short-acting β2 agonists (should not be used on more than 2 occasions in a week, excluding for prophylactic treatment).
* Subjects have no current exposure to allergens to which the subject experiences asthmatic responses (except for the house dust mite).
* Positive methacholine challenge (PC20 ≤16 mg/mL) at screening (Visit 2).
* Positive skin-prick test to at least one common aeroallergen at screening (Visit 1).
* Positive early and late airway responses during the screening allergen challenge. The EAR will be a fall in FEV1 of ≥20% during the 2 hours after allergen challenge. The LAR will be defined as a fall in FEV1 of ≥15% during the 3-7 hours after allergen challenge.
* Pre-bronchodilator FEV1 at screening (Visit 1) ≥70% of predicted normal value.

Weight

• Body mass index (BMI) within the range 18 to 35 kg/m2 (inclusive).

Sex • Male or female

Reproduction

* Negative serum pregnancy test for female subjects at Screening Visit 1.
* WOCBP should be stable on their chosen method of highly effective birth control for a minimum of 3 months prior to Visit 1, and willing to use this for the entire duration of the study (from the time they sign the ICF), and for 1 month after the last dose of study treatment. With the exception of abstinence, addition of a barrier method (such as a condom) must be used from Visit 1 until 1 month after the last dose of study treatment. Female subjects must not donate ova for the same time period
* Male subjects must be surgically sterile or using an acceptable method of contraception for the duration of the study (from the time they sign consent) and for 1 month after the last dose of study treatment to prevent pregnancy in a partner (unless the partner is considered postmenopausal). Male subjects must not donate or bank sperm during this same time period.

Additionally, for randomization into the study (baseline Visit 6), the subject must fulfil the following additional criteria:

* Negative urine pregnancy test for female subjects, confirmed pre dose prior to randomization.
* Visit 6 pre dose methacholine PC20 ≤1 doubling concentration lower than the corresponding baseline value at Visit 2.
* Ability to produce a sputum sample and viable cytospin for assessment of the cell differential count at the screening allergen challenge. The purpose of this analysis is to support exploratory endpoints only and is not related to treatment decisions.
* A Visit 6 pre-dose FEV1 that is not more than 10% lower than that measured at the screening Visit 2, to demonstrate asthma stability.

Exclusion criteria

Medical conditions

* A worsening of asthma or a respiratory tract infection from 6 weeks prior to Visit 1 or during the screening period, requiring a change of treatment.
* Any history of life-threatening asthma attack or asthma attack requiring admission to an intensive care unit and/or ventilation.
* A medical history or evidence of medical conditions which in the Investigator's opinion makes it undesirable for the subject to participate in the study, including but not limited to:

  1. lung disease (excluding sleep apnea) other than mild allergic asthma
  2. history of diabetes, metabolic syndrome, Gilbert syndrome, hepatic impairment, hypertriglyceridemia, or familial lipid disorders
  3. clinically significant hypotensive episodes or symptoms of fainting, dizziness, or light headedness
  4. cardiovascular disease, particularly coronary artery disease, hypertension, congestive heart failure or any clinically important abnormalities in rhythm, conduction or morphology of the ECG at rest that may interfere with the interpretation of QT interval corrected (QTc) interval changes.
  5. significant neurologic disease, including transient ischemic attack, stroke, or seizure disorder
  6. alcoholism, drug dependency or abuse
  7. latent or chronic infection (eg, recurrent sinusitis, genital or ocular herpes, urinary tract infection) or at risk of infection (eg, surgery) within 90 days of screening
  8. malignancy in the previous 5 years other than superficial basal cell carcinoma.
* Prolonged QT interval corrected using Fridericia's formula (QTcF) >450 milliseconds (ms) based on ECG (at Visit 1 or Visit 6 pre-dose) or family history of long QT syndrome
* Persistent or intermittent bundle branch block, intermittent second or third degree atrial ventricular (AV) block or AV dissociation (at Visit 1 or Visit 6).
* Current smokers. Ex-smokers must not have smoked or used nicotine or cannabis products (including e-cigarettes) for a minimum of 6 months prior to enrolment and should not have a smoking history ≥10 pack years.
* Excessive intake of caffeine-containing drinks or food (eg, coffee, tea, chocolate) as judged by the Investigator.

Prior/concomitant therapy

* Intention to use any concomitant medication that is not permitted or failure to undergo the required washout period for a prohibited medication.
* Chronic use of any other medication for treatment of allergic lung disease other than short acting β2-agonist.
* Subject who has a scheduled in-patient surgery or hospitalization during the study.
* Previous use of a mechanistic target of rapamycin (mTOR) antagonist (eg, rapamycin, everolimus) or PI3K inhibitor (selective or non-selective PI3K inhibitor).

Prior/concurrent clinical study experience

• Participation in another clinical study with an investigational product administered from 30 days (or 5 half lives) before Visit 1.

Note: refer to prohibited/restricted medications list for required washouts from previous investigational treatments.

* Subjects with a known hypersensitivity (as judged by the Investigator) to drugs with a similar class to AZD8154.
* Previously received AZD8154 or randomized to treatment in the present study.

Diagnostic assessments

* Clinically significant abnormalities in laboratory test results at Visit 1 or during the screening period as judged by the Investigator.
* Any values outside the normal range for the following parameters at Visit 1:

  1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level ≥1.5 times the upper limit of normal (ULN).
  2. Absolute neutrophil count ≤1.5 x 109/L.
* Positive serology at Visit 1 (HIV-1; HIV-2; Hepatitis B & C).
* Subjects with latent or active tuberculosis (TB), as confirmed by a positive QuantiFERON® - TB Gold test or as judged by the Investigator at Visit 1.

Note: subjects will be allowed to continue with screening and baseline assessments whilst the results are pending but must not be randomized into the study until the test results confirm the subject does not have TB.

Other exclusions

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff, staff at the study site, and other third party staff involved in the study).
* Judgement by the Investigator that the subject should not participate in the study if the subject is unlikely or unwilling to comply with study procedures, restrictions and requirements.
* Female subjects who are currently pregnant (confirmed with positive pregnancy test) or breast feeding or planning a pregnancy (also applies to male subjects), within the study period or 1 month following the last dose of study treatment.
* If a subject agrees to participate in the optional genetic research, the following exclusion criteria will apply:

  1. Previous allogeneic bone marrow transplant.
  2. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genomic sample collection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2021-11-10 (Estimated); Study Completion 2021-11-10 (Estimated)

PRIMARY OUTCOMES:
Maximal percentage decrease in forced expiratory volume in 1 second (FEV1) 3-7 hours post-allergen challenge | At day 9
  To evaluate the effect of AZD8154 on the allergen-induced late asthmatic response 3-7 hours post-allergen challenge (LAR3-7hr) when compared with placebo
Area under the curve (AUC) of time adjusted percent decrease in FEV1 in late asthmatic response (LAR) 3-7hr | At day 9
  To evaluate the effect of AZD8154 on the allergen-induced late asthmatic response 3-7 hours post-allergen challenge (LAR3-7hr) when compared with placebo

SECONDARY OUTCOMES:
Maximum percentage fall in FEV1 0-2 hours post-allergen challenge | At day 9
  To investigate the effect of AZD8154 compared with placebo by early asthmatic response (EAR0-2hr) by assessment of maximum percentage fall in FEV1 0-2 hours post-allergen challenge
AUC of time adjusted percent decrease in FEV1 curve in EAR0-2hr | At day 9
  To investigate the effect of AZD8154 compared with placebo by early asthmatic response (EAR0-2hr) by assessment of maximum percentage fall in FEV1 0-2 hours post-allergen challenge
PC20 dose of methacholine causing ≥20% fall in FEV1 | At Day 1, Day 8 and Day 10
  To evaluate airway hyperresponsiveness (AHR) at baseline, pre-allergen challenge and at 24 hours post-allergen challenge by assessment of methacholine PC20 (concentration of inhaled methacholine that produces a 20% fall in FEV1)
FENO at baseline, pre-allergen challenge and at 7 and 24 hours post-allergen challenge | At Day 1, Day 8, Day 9 and Day 10
  To assess changes in fractional exhaled nitric oxide (FENO) pre-allergen challenge and at 7 and 24 hours post-allergen challenge
Plasma concentrations of AZD8154 pre- and post-allergen challenge | At pre-dose on day 1, day 2 to day 7, 10 minutes post-dose on day 8 and pre-dose and 1, 2, 4 and 8 hours post-dose on day 9, pre-dose on day 10 and day 17 (follow-up)
  To investigate drug exposure of AZD8154 in subjects with mild allergic asthma
Number of subjects with adverse events or abnrmal finding in vital signs, pulse oximetry, electrocardiogram (ECG), clinical chemistry / haematology / urinalysis, physical examination and spirometry | Up to 9.5 weeks, from screening (45 days), treatment (7 days) to follow-up period (10 days)
  To evaluate the safety and tolerability of 10 days repeated dosing AZD8154 compared with placebo in subjects with mild allergic asthma

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Site, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home